CLINICAL TRIAL: NCT02624375
Title: Immune Response to Shingles Vaccination
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Christine Johnston, Associate Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00001399; 53354 (Other Grant/Funding Number: Merck)
Record Dates: First submitted 2015-12-02; First posted 2015-12-08 (Estimated); Results first posted 2019-12-05 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Shingles
MeSH Terms: conditions — Herpes Zoster | interventions — Herpes Zoster Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 10 persons over 70 years of age that received Zostavax (Experimental): 10 persons over 70 years of age that received Zostavax (single 0.65-mL dose subcutaneously in the deltoid region of the upper arm)
  Interventions: Drug: Zoster Vaccine Live

INTERVENTIONS:
Drug: Zoster Vaccine Live
  Other Names: ZOSTAVAX

SUMMARY:
The purpose of this study is to learn more about the immune response to varicella zoster virus (VZV).

DETAILED DESCRIPTION:
Participants 70 years of age or older will receive the FDA-approved shingles vaccine (Zostavax). Blood samples and optional skin biopsies will be obtained before and after vaccination to study the immune responses to shingles vaccination.

ELIGIBILITY:
Inclusion Criteria:

* 70 years of age or older.
* History of chickenpox.

Exclusion Criteria

* Previous vaccination with Zostavax or with the chickenpox vaccine.
* History of ever having had shingles.
* Been in close contact with a person who had chickenpox or shingles in the past 5 years.
* VZV seronegative
* Taking systemic suppressive regular doses of drugs with anti-VZV activity such as acyclovir, famciclovir, or valacyclovir. Episodic use is allowed. For Cohort 1: medication cannot be taken 24 hours prior to or 30 days after receiving Zostavax per CDC recommendations.
* HIV seropositive.
* Hepatitis C infection or active Hepatitis B infection.
* History of a life-threatening allergic reaction (anaphylactic/anaphylactoid reaction) to gelatin, neomycin, or any other component of shingles vaccine. Neomycin allergy manifested as contact dermatitis is not an exclusion.
* Has immunosuppression as a result of an underlying illness (e.g. leukemia, lymphoma or other malignant neoplasms) or treatment with immunosuppressive or cytotoxic drugs, or use of anticancer chemotherapy or radiation therapy.
* Has long-term use of oral or parenteral steroids (>7 days), or high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding 6 months (nasal and topical steroids are allowed).
* Women of child-bearing potential only: pregnant or planning to become pregnant 3 months post vaccination
* Donated blood in the past 8 weeks or planning to donate blood during the study
* Weighs less than 110 lbs
* Has any condition or medical history that would, in the opinion of the site principal investigator place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Additional exclusions for optional skin biopsy:

1. Has an acute or chronic medical condition that, in the opinion of the investigator, would render biopsies unsafe
2. History of coagulopathy or taking medication that may cause bleeding (long term aspirin, heparin, coumadin)
3. History of keloid formation or excessive scarring
4. History of frequent cellulitis or boils (>3 episodes in past 2 years) requiring antibiotic therapy.
5. Allergy to lidocaine, silver nitrate, or mupirocin.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Washington Virology Research Clinic, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from September 2016 to January 2018. Recruitment was done by placing flyers at retirement homes and by contacting persons over 70 who had previously been enrolled in research studies including giving informed written consent to be re contacted for future studies.
Groups:
- Persons 70 and Over Receiving Zostavax (Zoster Vaccine Live): We administered Zostavax at the FDA approved dose and route to an FDA-indication-approved population, namely healthy adults 70 and over. We administered vaccine to 10 persons as proposed in the protocol.
Period: Overall Study
Arm/Group | Persons 70 and Over Receiving Zostavax (Zoster Vaccine Live)
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Person 70 and over receiving Zostavax
Arm/Group | Persons 70 and Over Receiving Zostavax (Zoster Vaccine Live)
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 74.5 [70 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
no history of shingles or shingles vaccination [Count of Participants; unit: Participants] | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Th1 Cytokine Positive VZV-specific CD4 T-cells in Blood
Description: To determine if Zostavax, when given as FDA indicated, boosts VZV-specific T-cells in the blood
Time Frame: 6 months
Population: 10 persons 70 and older who received Zostavax
Measure: Median (Inter-Quartile Range); unit: percentage of CD4 T cells
Arm/Group | Persons 70 and Over Receiving Zostavax (Zoster Vaccine Live)
Number analyzed (Participants) | 10
percentage of CD4 T cells | 0.02 [0 to 0.07]

2. Primary Outcome: Percentage of Th1 Cytokine Positive VZV-specific CD4 T-cells in Skin
Description: To determine if shingles disease boosts the local level of VZV-specific T cells in skin 4 weeks after Zostavax
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: Percentage of CD4 T cells
Arm/Group | Persons 70 and Over Receiving Zostavax (Zoster Vaccine Live)
Number analyzed (Participants) | 10
Percentage of CD4 T cells | 0 [0 to 0.05]

3. Secondary Outcome: Number of Participants With Adverse Events Due to Zostavax
Description: To measure the occurrence of adverse events after Zostavax.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Persons 70 and Over Receiving Zostavax (Zoster Vaccine Live)
Number analyzed (Participants) | 10
Participants | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Persons 70 and Over Receiving Zostavax (Zoster Vaccine Live)
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-16): https://cdn.clinicaltrials.gov/large-docs/75/NCT02624375/Prot_SAP_000.pdf